CLINICAL TRIAL: NCT01237197
Title: Exenatide in Extreme Pediatric Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1009M88952
Record Dates: First submitted 2010-11-01; First posted 2010-11-09 (Estimated); Results first posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Exenatide; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exenatide, then Open-Label Exenatide (Experimental): Exenatide 5 micrograms (mcg): administered with injection twice per day (BID) for one month; up-titrated to 10 mcg twice per day for remainder of study (5 months)
  Interventions: Drug: Exenatide
- Placebo, then Open Label Exenatide (Placebo Comparator): Placebo injection twice a day for three months; Exenatide open label 5mcg twice a day for one month and up-titrated to 10mcg twice a day for remaining two months of study.
  Interventions: Drug: Exenatide; Drug: Placebo

INTERVENTIONS:
Drug: Exenatide — Exenatide 5 micrograms (mcg) twice per day (BID) for one month; up-titrated to 10 mcg twice per day for remainder of study.
  Other Names: Byetta
Drug: Placebo — Participants were randomized to a placebo injection for the first three months, then given open-label Exenatide for the remaining three months (Initiated at 5 mcg, twice per day, delivered by subcutaneous injection. After 1 month, exenatide was uptitrated to 10 mcg, twice per day for the remaining 2 months of the drug treatment phase).
  Other Names: Sugar pill
  Arms: Placebo, then Open Label Exenatide

SUMMARY:
Extreme pediatric obesity, the fastest growing category of obesity in youth, is associated with high risk for developing cardiovascular disease (CVD) and type 2 diabetes (T2DM). Obesity tracks strongly into adulthood and interventions early in life may reduce risk for developing cardiovascular disease and type 2 diabetes. Few drug therapies for weight loss have been evaluated in adolescents. Since exenatide is associated with weight loss and improves risk factors for cardiovascular disease and type 2 diabetes in adults, it may be useful in extremely obese youth. Our primary objective in this study is to generate preliminary data on the ability of exenatide to reduce body mass index (BMI) and improve risk factors for cardiovascular disease and type 2 diabetes in 26 extremely obese adolescents (age 12-19 years) in a three-month, randomized, double-blind, placebo-controlled pilot clinical trial. GLP-1 therapy has never been evaluated as a treatment for pediatric obesity and is an innovative approach to a challenging and significant health care problem.

DETAILED DESCRIPTION:
26 (approximately 13 per site) extremely obese (Body mass index [BMI] > or = 1.2 times the 95th percentile or BMI > or = 35 kg/m2) adolescents (age 12-19 years old) will be enrolled in a six-month study consisting of a three-month, randomized, double-blind (participants and investigators), placebo-controlled pilot clinical trial phase followed by a three-month open-label extension during which all participants will receive exenatide. For the initial three-month phase, participants will be equally (by site) and randomly assigned to one of two groups: 1) exenatide plus lifestyle modification, or 2) placebo plus lifestyle modification. Following baseline testing, subjects will be randomly assigned to study group. Participants will return at one-month for titration and assessment of safety (blood draw and adverse event assessment) and injection/lifestyle modification compliance and at three-months for reassessment of baseline variables and injection/lifestyle modification compliance and allocation to study drug for the three-month open-label extension. Participants will return at four-months for assessment of safety (blood draw and adverse event assessment) and injection/lifestyle modification compliance and at six-months for reassessment of baseline variables and injection/lifestyle modification compliance.

All subjects, regardless of group assignment, will participate in the clinical lifestyle modification program offered through either the University of Minnesota or Children's Hospitals and Clinics weight management programs. Participants and their families receive regular (approximately bi-monthly) face-to-face and/or phone behavioral-, dietary-, and physical activity-counseling from a multi-disciplinary team of health care professionals including physicians, dieticians, registered nurses, psychologists, and exercise physiologists.

Screening will include review of medical records for previous clinical and laboratory data. The following measures will be collected at baseline, 3 months, and 6 months. Subject will be asked to fast for a minimum of 12 hours.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index > or = 1.2 times the 95th percentile (based on gender and age) or Body mass index > or = 35 kg/m2
* 12-19 years old

Exclusion Criteria:

* Type 1 or 2 diabetes mellitus
* Previous (within 3-months) or current use of weight loss medication (patients may undergo washout)
* Previous bariatric surgery
* Recent initiation (within 1-month) of anti-hypertensive or lipid medication
* Previous (within 1-month) or current use of medication to treat insulin resistance or hyperglycemia (patients may undergo washout)
* Major psychiatric disorder
* Pregnant or planning to become pregnant
* Tobacco use
* Liver/renal dysfunction
* History of pancreatitis
* Obesity associated with genetic disorder
* Hyperthyroidism or uncontrolled hypothyroidism
* Uncontrolled hypertriglyceridemia (=300 mg/dL)
* Current eating disorder
* Previous (within 3-months) or current use of drugs associated with weight gain (e.g. steroids/anti-psychotics)

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2010-10; Primary Completion 2012-05 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron S. Kelly, Ph.D., Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - Children's Hospitals and Clinics of Minnesota, Saint Paul, Minnesota

REFERENCES:
- [Derived] Kelly AS, Rudser KD, Nathan BM, Fox CK, Metzig AM, Coombes BJ, Fitch AK, Bomberg EM, Abuzzahab MJ. The effect of glucagon-like peptide-1 receptor agonist therapy on body mass index in adolescents with severe obesity: a randomized, placebo-controlled, clinical trial. JAMA Pediatr. 2013 Apr;167(4):355-60. doi: 10.1001/jamapediatrics.2013.1045. PMID 23380890

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the University of Minnesota, Amplatz Children's Hospital Pediatric Weight Management Clinic in Minneapolis or the McNeely Pediatric Diabetes Center and Endocrinology Clinic, Children's Hospitals and Clinics of Minnesota in St Paul.
Groups:
- Exenatide: Exenatide 5 micrograms (mcg): administered with injection twice per day (BID) for one month; up-titrated to 10 mcg twice per day for remainder of study (5 months)
  Open label Exenatide : Exenatide 5 micrograms (mcg) twice per day (BID) for one month; up-titrated to 10 mcg twice per day for remainder of study.
- Placebo Injection: Placebo injection twice a day for three months; Exenatide open label 5mcg twice a day for one month and up-titrated to 10mcg twice a day for remaining two months of study.
  Open label Exenatide : Exenatide 5 micrograms (mcg) twice per day (BID) for one month; up-titrated to 10 mcg twice per day for remainder of study.
Period: Randomization Period
Arm/Group | Exenatide | Placebo Injection
Started | 13 | 13
Completed | 12 | 10
Not Completed | 1 | 3
Period: Open Label Period
Arm/Group | Exenatide | Placebo Injection
Started | 12 | 10
Completed | 12 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide | Placebo Injection | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 13 | 26
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.9 (1.76) | 15.5 (1.88) | 15.2 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Body Mass Index at 3-months
Description: As results are measured by BMI reduction, percent change (reduction) in BMI is primary outcome measure.
Time Frame: Baseline and 3-months
Measure: Mean (Standard Deviation); unit: percentage of change in BMI
Groups:
- Exenatide: Exenatide 5 micrograms (mcg): administered with injection twice per day for one month; up-titrated to 10 mcg twice per day for remainder of study (5 months)
  Open Label Exenatide : Exenatide 5 micrograms (mcg) twice per day for one month; up-titrated to 10 mcg twice per day for remainder of study.
- Placebo Injection: Placebo injection twice a day for three months; Exenatide open label 5mcg twice a day for one month and up-titrated to 10mcg twice a day for remaining two months of study.
  Open Label Exenatide : Exenatide 5 micrograms (mcg) twice per day for one month; up-titrated to 10 mcg twice per day for remainder of study.
Arm/Group | Exenatide | Placebo Injection
Number analyzed (Participants) | 12 | 10
percentage of change in BMI | -2.9 (1.8) [-5.02 to -0.37] | -0.15 (3.2)

ADVERSE EVENTS:
Arm/Group | Exenatide | Placebo Injection
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 12/13 | 12/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exenatide (N=13) | Placebo Injection (N=13)
Nausea (Gastrointestinal disorders) | 8 (13) | 4 (4)
Vomiting (Gastrointestinal disorders) | 4 (5) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 4 (4)
Headache (Nervous system disorders) | 3 (4) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No